CLINICAL TRIAL: NCT03610685
Title: Persistence of Inflammation and Study of T2 Pathways Following Inhibition of InterLeukin-5 With Mepolizumab in Severe Eosinophilic Asthma
Brief Title: Inflammation Following Mepolizumab and Oral Corticosteroids in Asthma
Acronym: MAPLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: GN17RM707
Record Dates: First submitted 2018-03-27; First posted 2018-08-01 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: Severe asthma; Mepolizumab; IL5; Steroid resistance; Eosinophilic asthma; Type 2 inflammation
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will be given 2 weeks of placebo treatment. The placebo capsules will be taken once a day orally. The daily dose of placebo treatment will match the Prednisone dose for each participant.
  Interventions: Drug: Placebo oral capsule
- Prednisolone (Active Comparator): Participants will be given 2 weeks of prednisolone treatment. This is administered orally once a day. The daily dose is calculated according to 0.5mg/kg with a maximum dose of 40mg per day.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Given daily for 2 weeks
  Arms: Prednisolone
Drug: Placebo oral capsule — Given daily for 2 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The aim of the project is to study the persistence of inflammation after addition of an interleukin-5 (IL-5) blocker in severe eosinophilic asthma as a study of untreated pathways in these patients.

DETAILED DESCRIPTION:
Mepolizumab, a humanized monoclonal antibody (mAb) antagonizes IL-5 and through a selective inhibition of eosinophilic inflammation, reduces the number of eosinophils in sputum and blood, leading to a reduction in asthma exacerbations and a need for systemic glucocorticoids. Once this therapy has been initiated for severe eosinophilic asthma, the additional role of oral corticosteroids is questionable as their main target is reduction of eosinophils and hence responsiveness to oral corticosteroids in patients in a stable state of asthma may reduce.

Using two weeks of high dose prednisolone versus placebo in a crossover design after 12 weeks of mepolizumab therapy will allow an understanding of the pathways that remain steroid responsive following IL-5 suppression.

This is an exploratory study with no single primary end point. The objective of the study is to assess the change in airway inflammation following oral corticosteroids versus placebo and the airway inflammation while on mepolizumab in stable state of asthma.

Note: Mepolizumab is not an intervention in this study; it is initiated as part of usual NHS care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years at consent.
* Able and willing to provide written informed consent and to comply with the study protocol.
* Severe asthma diagnosis confirmed after assessment by an asthma specialist.
* Suitable for mepolizumab as per NICE/SMC Clinical Guidelines.

Exclusion Criteria:

* Maintenance oral corticosteroid treatment within the past four weeks.
* Acute exacerbation requiring oral corticosteroids in the four weeks prior to consent.
* Other clinically significant medical disease or uncontrolled concomitant disease despite treatment that is likely, in the opinion of the investigator, to require a change in therapy or impact the ability to participate in the study or be significantly worsened by oral corticosteroids.
* History of current alcohol, drug, or chemical abuse or past abuse that would impair or risk the subject's full participation in the study, in the opinion of the investigator.
* Treatment with an investigational agent within 30 days of Visit 1 (or five half-lives of the investigational agent, whichever is longer).
* Women of child-bearing potential who are pregnant, lactating, planning pregnancy during the study period or are unwilling to use a highly effective form of contraception.
* Known hypersensitivity to prednisolone or its excipients.
* Previous psychiatric adverse reactions to steroid therapy in the past.
* Concomitant medication with systemic anti-fungals such as ketoconazole, retinoids, tetracycline, other systemic immunosuppressants e.g. ciclosporin, azathioprine, mycophenolate and live vaccines during the crossover trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Change in exhaled nitric oxide measured in parts per billion | Through study completion, an average 20 weeks.
  Measured at study visits using a Niox machine.
Change in sputum differential cell counts measured in absolute cell count. | Through study completion, an average 20 weeks
  Induced sputum

OTHER OUTCOMES:
Change in asthma control and quality of life questionnaires | Through study completion, an average 20 weeks.
  Asthma control questionnaire includes 5 questions related to asthma control. Each question is scored from 0 to 6 with the highest number representing poorer outcome / asthma control.
  Asthma quality of life questionnaire includes 32 questions related to quality of life. Each question is scored from 1 to 7 with the highest number representing better outcome / quality of life.
Change in visual asthma symptom scores | Through study completion, an average 20 weeks
  Symptoms visual analogue scale asks 3 questions related to asthma control. A
Oscillometry | Through study completion, an average 20 weeks
  For small airway function to correlate with inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Chaudhuri, MD, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Asthma and copd research centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided